CLINICAL TRIAL: NCT03729505
Title: Impact of Pyloric Injection With Magnesium Sulphate and Lidocaine Mixture on Early Postoperative Outcome After Laparoscopic Sleeve Gastrectomy
Brief Title: Impact of Pyloric Injection of Magnesium Sulfate and Lidocaine Mixture on Outcome After Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura66
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyloric injection of magnesium sulfate and lidocaine mixture (Active Comparator): After sleeve gastrectomy, the pylorus is injected with a mixture of magnesium sulfate and lidocaine
  Interventions: Procedure: Pyloric injection of magnesium sulfate and lidocaine mixture
- Pyloric injection of saline (Active Comparator): After sleeve gastrectomy, the pylorus is injected with normal saline
  Interventions: Procedure: Pyloric injection of saline

INTERVENTIONS:
Procedure: Pyloric injection of magnesium sulfate and lidocaine mixture — 100 mg / 2 ml of magnesium sulphate (Magnesium Sulfate®) is mixed with 5 ml of 2% lidocaine and injected in the pylorus
  Arms: Pyloric injection of magnesium sulfate and lidocaine mixture
Procedure: Pyloric injection of saline — 5 ml of normal saline is injected in the pylorus
  Arms: Pyloric injection of saline

SUMMARY:
Postoperative nausea and vomiting is a common adverse effect after sleeve gastrectomy, mostly due to increased intragastric pressure. The present trial aimed to assess the effect of pyloric injection of mixture of magnesium sulfate and lidocaine on postoperative gastric intraluminal pressure and incidence of nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients that aged between18 and 65 years.
* American Society of Anesthesiologists (ASA) class I - III.
* Morbidly-obese patients who failed to achieve and maintain a clinically significant weight loss through supervised non-surgical methods for at least 6 months.
* Surgery was conducted as the first line of treatment in case of patients with BMI ≥ 50 kg/m2 (super obese).

Exclusion Criteria:

* Obesity secondary to endocrine disorders.
* History of any previous bariatric procedure.
* Impaired intellectual capacity or major psyciatric disorder.
* Sweet eaters who would not adopt a change of postoperative eating habits.
* Lack of willingness and motivation to embrace postoperative lifestyle changes.
* Substance abuse.
* Pregnancy or expected pregnancy in the following 12 to 18 months.
* Severe gastroesophageal reflux disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | first 24 hours after surgery
  incidence of postoperative nausea and vomiting as measured by special impact scale

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided